CLINICAL TRIAL: NCT00944463
Title: Randomized Double-blinded, Placebo-controlled Phase II Trial of Simvastatin and Gemcitabine in Advanced Pancreatic Cancer Patients
Brief Title: Trial of Simvastatin and Gemcitabine in Pancreatic Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Suk Park, professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-07-065
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: advanced pancreatic cancer; gemcitabine; simvastatin; placebo
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine+simvastatin (Experimental): Gemcitabine and simvastatin
  Interventions: Drug: Gemcitabine+simvastatin
- Gemcitabine+Placebo (Placebo Comparator): Gemcitabine plus Placebo
  Interventions: Drug: Gemcitabine+Placebo

INTERVENTIONS:
Drug: Gemcitabine+simvastatin — Gemcitabine and simvastatin
  Other Names: Gemcitabine and simvastatin
  Arms: Gemcitabine+simvastatin
Drug: Gemcitabine+Placebo — Gemcitabine plus Placebo
  Other Names: Gemcitabine plus Placebo
  Arms: Gemcitabine+Placebo

SUMMARY:
The purpose of this study is to determine whether simvastatin is effective in the treatment of advanced pancreatic cancer patients.

DETAILED DESCRIPTION:
Randomized double-blinded, placebo-controlled phase II trial of simvastatin and gemcitabine in advanced pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Histologically or cytologically confirmed, metastatic or unresectable pancreatic adenocarcinoma (if repeated biopsy (>3) fails or if biopsy is not feasible, the inclusion of the patient will be determined by the central PI)
3. ECOG performance status of 0~2
4. no radiotherapy within 1 month of the study entry
5. measurable or evaluable lesion according to RECIST criteria
6. no prior history of chemotherapy for pancreatic cancer (gemcitabine-based adjuvant chemotherapy ≥ 12 months from the study entry will be allowed)
7. adequate marrow, hepatic, renal and cardiac functions (absolute neutrophil count ≥ 1.5 x 109/L; platelet count ≥ 75 x 109/L, serum creatinine ≤ 1.5 x ULN), serum aspartate aminotransferase/alanine aminotransferase ≤ 5 x ULN or ≤ 10 x ULN if liver abnormalities are due to underlying malignancy; total bilirubin ≤ 2.0 x ULN
8. written informed consent must be provided

Exclusion Criteria:

1. severe co-morbid illness and/or active infections
2. pregnant or lactating women
3. active CNS metastases not controllable with radiotherapy or corticosteroids A.patients with symptoms suggestive of CNS metastases must undergo radiologic evaluation to rule out metastases B.patients with known, asymptomatic CNS lesions are permitted
4. known history of hypersensitivity to study drugs
5. patients who are currently on statin therapy or has taken statin as lipid lowering agents within 1 year of the study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Time to progression | Every 2 cycles until progression

SECONDARY OUTCOMES:
Safety profiles of gemcitabine/simvastatin | Every cycle until progression
Response rate | Every 2 cycles until progression
Duration of response | Every 2 cycles until progression
Overall survival | Every 3 months
Correlative analyses | after completion of accrual

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, M.D.,Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea